CLINICAL TRIAL: NCT01467609
Title: PillCam Colon Capsule Endoscopy Versus Conventional Colonoscopy for the Detection of the Severity and Extent of Ulcerative Colitis
Brief Title: PillCam Colon Capsule Endoscopy for Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjyyxhk2319
Record Dates: First submitted 2011-10-20; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Ulcerative Colitis
Keywords: Pillcam colon capsule endoscopy; conventional colonoscopy; ulcerative colitis; endoscopic manifestation; colonoscopy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — regular biopsy was taken during conventional colonoscopy according to the activity and position of ulcerative colitis involved.
Oversight: Data Monitoring Committee: No

SUMMARY:
Pillcam colon capsule (PCC) endoscopy is a novel strategy tool to inspect colon mucosa. The aim of the present study is to evaluate if PCC endoscopy is able to precisely investigate patients with ulcerative colitis and reach high consistency to conventional colonoscopy.

DETAILED DESCRIPTION:
Symptomatic patients with confirmed ulcerative colitis (UC) were enrolled in this prospective single-center study. No sooner had patients gone through Pillcam colon capsule (PCC) endoscopy solution than they got conventional colonoscopy which is recognized as the "gold standard" examination technique. The extent of mucosal damage and inflammatory lesions during both modalities were recorded for comparison. In addition, the regimen of bowel preparation, completion rate, colonic cleanliness, compliance or adverse events were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-70)
* Ulcerative Colitis history
* Suffering from symptoms such as hematochezia, diarrhea or abdominal pain

Exclusion Criteria:

* Patients with a high risk for capsule retention (such as intestinal diverticula, acute abdominal pain without regular defecation indicating intestinal obstruction or a history of abdominal operation or intestinal reconstructed operation),
* Patients allergic to sodium phosphate or polyethylene glycol (PEG) solution,
* Patients with a history of Crohn's disease
* Patients with serious systematic diseases such as congestive heart failure, renal failure or severe liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: academic hospital endoscopist of digestive department
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the accuracy of PCC endoscopy in the survey of ulcerative colitis compared with conventional compared with conventional
  the severity of patients investigated by PCC endoscopy and conventional colonoscopy the extent of evolved lesions extent investigated by PCC endoscopy and conventional colonoscopy the safety of PCC endoscopy course (eg: adverse events during bowel preparation and the course; the completion rate)

SECONDARY OUTCOMES:
the gastrointestinal transit time (transit time from ingestion to excretion), cecum arrival time (transit time from ingestion to the cecum), and colon residence time (transit time from the arrival in the cecum to excretion)
clinical data such as age, gender,chief complaint
the Mayo score of each case
the quality of colonic preparation
  4 grades contain excellent, good, fair and poor

CONTACTS AND LOCATIONS:
Overall Officials: zhi zheng Ge, MD. Ph.D, Principal Investigator — Clinical Professor of Gastroenterology Department, Shanghai Renji Hospital; Director, Head of Digestive Endoscopy Department, Shanghai Renji Hospital